CLINICAL TRIAL: NCT01350427
Title: Effects of Leucine, Branched-chain Amino Acids, and Resistance Exercise on Skeletal Muscle Remodelling Signaling Pathways: a Randomized, Double-blind, and Placebo-controlled Study
Brief Title: Branched-chain Amino Acids, and Resistance Exercise on Skeletal Muscle Signaling Pathways
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Humberto Nicastro, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2011/04690-6
Record Dates: First submitted 2011-05-02; First posted 2011-05-09 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Healthy
Keywords: leucine supplementation; BCCA supplementation; resistance exercise-induced muscle remodeling

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Leucine (Experimental)
  Interventions: Dietary Supplement: Leucine supplementation
- BCAA (Experimental)
  Interventions: Dietary Supplement: BCAA supplementation
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Alanine supplementation

INTERVENTIONS:
Dietary Supplement: Leucine supplementation — 1 bout of resistance exercise and supplementation of 4.0 g of leucine + 5.6 g of alanine
  Arms: Leucine
Dietary Supplement: BCAA supplementation — 1 bout of resistance exercise and supplementation of 4.0 g of leucine + 2.8 g of isoleucine + 2.8 g of valine
  Arms: BCAA
Dietary Supplement: Alanine supplementation — 1 bout of resistance exercise and supplementation of 9.6 g of alanine
  Arms: Placebo

SUMMARY:
This study aims to evaluate the effects of leucine and branched-chain amino acids supplementation on skeletal muscle remodeling signaling pathways induced by resistance exercise.

ELIGIBILITY:
Inclusion Criteria:

* Sedentaries
* Must be able to exercise
* Must be able to swallow tablets

Exclusion Criteria:

* Use of nutritional supplements
* Use of anti-inflammatory drugs

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2011-08; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Protein synthesis | 1 hour
  Phosphorylation of proteins involved in protein synthesis
Protein degradation | 1 hour
  Expression of protein involved in proteolytic pathway
Inflammation | 1 hour
  Expression of systemic and muscular cytokines

CONTACTS AND LOCATIONS:
Overall Officials: Claudia R da Luz, Master Student, Principal Investigator — University of Sao Paulo
Locations (1):
- University of São Paulo - School of Physical Education and Sports, São Paulo, São Paulo, Brazil